CLINICAL TRIAL: NCT05250726
Title: Evaluation of the Treatment of Symptomatic Scaphotrapeziotrapezoidal (STT) Osteoarthritis with a Treated, Devitalized and Sterile Meniscus Segment (MENISC-T) Placed in Joint Interposition
Brief Title: Use of a Treated, Devitalized and Sterile Meniscus Segment (MENISC-T) in the Treatment of Scaphotrapeziotrapezoid Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TBF Genie Tissulaire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MENISC-T-STT; 2020-A02916-33 (Other: IDRCB)
Record Dates: First submitted 2022-02-10; First posted 2022-02-22 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis Hand
Keywords: ScaphoTrapezioTrapezoid OsteoArthritis (STT OA)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MENISC-T (Experimental): Segmented, devitalized and sterile meniscus graft
  Interventions: Biological: MENISC-T

INTERVENTIONS:
Biological: MENISC-T — Decellularized, viro-inactivated, freeze-dried and sterile allogeneic graft of meniscus used as interposition at the STT joint

SUMMARY:
The purpose of this open, prospective and multi center trial is to evaluate the use of a treated, devitalized and sterile meniscus implant placed in joint interposition in the treatment of STT osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female; age between 18 and 75 years.
* Patient with symptomatic STT OA.
* Patient treated medically for functional signs for more than 3 months, without improvement, justifying a surgical intervention.
* Patient with a QuickDash score > 33 points (converted to 50%).
* Patient with wrist pain (VAS) in front of the STT joint at rest > 4/10.
* Patient who received the study information and provided consent.
* Member or beneficiary of a national health insurance plan.

Exclusion Criteria:

* Pregnant or breastfeeding woman; woman without effective contraception.
* Patient with functional rhizarthrosis that has not been stabilized or treated medically or surgically.
* Patient with signs of neuropathy with functional disorders such as hyperesthesia.
* Patient with uncontrolled epilepsy or neuropathy that contraindicates locoregional anesthesia.
* Person confined by a judicial or administrative decision.
* Adult subjected to legal protection measures or unable to provide his/her consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Decrease of the symptomatology related to the STT OA | 12 months
  Quality of life related to STT OA evaluated using Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire (0 = no disability, 100 = most severe disability); a decrease of 25% of the score is expected between subject's inclusion and the 12-month postoperative visit

SECONDARY OUTCOMES:
Absence of toxicity | Through study completion - average of 12 months
  Absence of adverse events
Increase of thumb strength | 1 month, 3 months, 6 months, 12 months
  Thumb strength measured in kg by two-point pinch strength test
Decrease of pain related to STT OA | 1 month, 3 months, 6 months, 12 months
  Pain evaluated from 0: no pain to 10: worst imaginable pain on visual analog scale (VAS)
No apparent anomaly of joint space | 12 months
  Joint space evaluated on radiography using Crosby's classification

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Chirurgical de la Main et du Membre Supérieur, Villeurbanne, France